CLINICAL TRIAL: NCT02626728
Title: A Prospective Quality Assurance Feasibility Study of Laparoscopic Assisted Transanal Minimally Invasive Surgery (TAMIS) for Rectal Cancer
Brief Title: A Prospective Feasibility Study for TAMIS
Acronym: TAMIS
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, M.D, PhD, Hvidovre University Hospital
Other Study IDs: 123-TAMIS
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Transanal Endoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laparoscopic assisted transanal surgery (TAMIS) — all patients included recieve laparoscopic assisted transanal minimally invasive surgery

SUMMARY:
Most recently, the Transanal Minimally Invasive Surgery (TAMIS) approach combined with single-port technology has allowed that pelvic surgery can be laparoendocopically performed from both its abdominal and perineal aspects.Previously, a strong negative association between medium- and long-term survival and male gender with narrow pelvis have been reported. TAMIS has a significant potantial for improving the quality of the surgical resection of rectal tumors in men with visceral obesity and narrow pelvis. This group of patients have also a high rate of conversion to open surgery. Focusing on improvement in intraoperative conditions and surgical techniques rather than routine conventional procedures may be the way to go concerning favorable short- and long-term outcomes. The selection of adequate surgical approach to the high-risk patients with visceral obesity and a bulky mesentery may prevent or limit the risk for anastomotic leakage and improve oncologic margin clearence. This is a prospective observational feasability study of the TAMIS-procedure.

ELIGIBILITY:
Inclusion criteria:

* rectal cancer with histological diagnosis
* tumors located between 10 - 4 cm from the anal verge measured with a rigid rectoscope.
* suitable for elective resection

exclusion criteria:

* preoperative magnetic resonance imaging (MRI) showing diameter of tumor size >6 cm
* American Society of Anesthesiologists (ASA) class IV and V
* anticipated need of intensive care unit (ICU)
* history of previous major abdominal surgery
* computer assisted tomography (CT) or MRI evidence of tumor infiltration of adjacent organs
* obese patient with body mass index >35kg/m2
* those, who do not understand the requirements of the protocol
* pregnancy
* more than one colorectal tumor

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a solitary rectal cancer, who is eligible for surgery. Patients with rectal cancer (T1-3 stages verified by MRI), regardless regional lymph-node status and distant metastasis, will be offered the operative procedure with TAMIS technique.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
morbidity | 30-days
  Clavien-Dindo

SECONDARY OUTCOMES:
mortality | 30-days
  death within 30-days
short-term oncological result | 30-days
  cancer-free resection margins

CONTACTS AND LOCATIONS:
Overall Officials: Mette W Christoffersen, M.D, PhD, Study Chair — Hvidovre Hospital University of Copenhagen
Locations (1):
- Hvidovre Hospital University of Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No